CLINICAL TRIAL: NCT03469544
Title: Long Non Coding RNA HOTAIR and Midkine as Biomarkers in Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saleh Abdelghafour, principle investigator, Assiut University
Other Study IDs: LNCRHAMBTC
Record Dates: First submitted 2018-03-10; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Creatinine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 (30): Patient with cancer thyroid proved by cytological analysis Interventions;complete blood picture ,serum urea and creatinine,liver function test,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body .
  specific test is quantitation of long non coding RNA HOTAIR by Real time polymerase chain reaction in peripheral blood ,Enzyme linked Immunosorbent Assay for serum midkine level
  Interventions: Other: complete blood picture ,serum urea and creatinine,liver function test,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body specific test Real time polymerase chain reaction
- Group 2 (30): Patient with benign thyroid nodule Interventions;complete blood picture ,serum urea and creatinine,liver function test ,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body .
  specific test is quantitation of long non coding RNA HOTAIR by Real time polymerase chain reaction in peripheral blood,Enzyme linked Immunosorbent Assay for serum midkine level
  Interventions: Other: complete blood picture ,serum urea and creatinine,liver function test,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body specific test Real time polymerase chain reaction
- Group 3 (30): Normal healthy subjects as control group Interventions;complete blood picture ,serum urea and creatinine,liver function test,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body .
  specific test is quantitation of long non coding RNA HOTAIR by Real time polymerase chain reaction in peripheral blood,Enzyme linked Immunosorbent Assay for serum midkine level
  Interventions: Other: complete blood picture ,serum urea and creatinine,liver function test,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body specific test Real time polymerase chain reaction

INTERVENTIONS:
Other: complete blood picture ,serum urea and creatinine,liver function test,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body specific test Real time polymerase chain reaction — complete blood picture ,serum urea and creatinine,liver function test,T3,T4,thyroid stimulating hormone,thyroglobuline and thyroglobuline anti body .
  specific test is quantitation of long non coding RNA HOTAIR by Real time polymerase chain reaction in peripheral blood,Enzyme linked Immunosorbent Assay for serum midkine level

SUMMARY:
Thyroid cancer is the most prevalent endocrine malignancy.Papillary thyroid carcinomas and follicular thyroid carcinomas account for 95% of all thyroid cancer cases. They are clinically classified as well-differentiated thyroid carcinomas due to their biological behavior resembling normal follicular cells and good responsiveness to surgery and radioiodine therapy . However, they are usually curable when discovered at early stages, but survival rates may be reduced from 100% in stages I and II to 50% at stage IV So,early detection is the key for successful treatment and reduction of mortality.

pathological analysis by fine-needle aspiration biopsies has some limitations including difficulty in sampling small tumors, inconclusive diagnosis in up to 35% of patients and bleeding. Thus, biomarkers for diagnosis are needed.

DETAILED DESCRIPTION:
Thyroid cancer is the most prevalent endocrine malignancy.Papillary thyroid carcinomas and follicular thyroid carcinomas account for 95% of all thyroid cancer cases. They are clinically classified as well-differentiated thyroid carcinomas due to their biological behavior resembling normal follicular cells and good responsiveness to surgery and radioiodine therapy . However, they are usually curable when discovered at early stages, but survival rates may be reduced from 100% in stages I and II to 50% at stage IV So,early detection is the key for successful treatment and reduction of mortality.

pathological analysis by fine-needle aspiration biopsies has some limitations including difficulty in sampling small tumors, inconclusive diagnosis in up to 35% of patients and bleeding. Thus, biomarkers for diagnosis are needed.

The concept of liquid biopsy was proposed in contrast to the traditional tissue biopsy which is particularly important for solid tumor diagnosis. It refers to the process of detecting genetic materials, using non-invasive method from blood or other body fluids.Long noncoding RNAs (LncRNAs) have recently been demonstrated to participate in cancer progression.HOTAIR is the type of non coding RNA that will be investigated for its ability to differentiate benign from malignant thyroid nodule Midkine a basic heparin-binding growth factor of low molecular weight, capable of exerting activities such as cell proliferation, cell migration, angiogenesis and fibrinolysis. Midkine expression is closely related with progression of tumor stage. If tumor tissues increase secretion of midkine, it becomes evident in serum.The expression of midkine gene in human tumor cells may reflect tumor formation and give clues to the biological behavior of neoplasms. Hence, the expression of midkine may serve as a tumor marker for diagnosis and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patient with thyroid mass

Exclusion Criteria:

* no other known organ malignancy no previous chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group(1) patient with thyroid cancer (30) Group(2) patient with begnin thyroid nodule (30) Group(3) normal healthy subjects as control (30)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-03-29 (Estimated); Primary Completion 2019-12-29 (Estimated); Study Completion 2020-03-29 (Estimated)

PRIMARY OUTCOMES:
Expression of long non coding RNA HOTAIR | 3 days
  Quantitation of long non coding RNA HOTAIR by real time polymerase chain reaction in peripheral blood

SECONDARY OUTCOMES:
level of serum midkine in thyroid cancer | 3 days
  Enzyme linked immunosorbent assay for estimation of serum midkine level

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aizizi Abudoureyimu*, Reyihanguli Maimaiti*, Sailike Magaoweiya, Duman Bagedati, Hao WenIdentification of long non-coding RNA expression profile in tissue and serum of papillary thyroid carcinoma Department of Vascular Thyroid Surgery, Gastrointestinal Vascular Center, The First Affiliated Hospital of Xinjiang Medical University, Urumqi 830054, Xinjiang, China.Int J Clin Exp Pathol 2016;9(2):1177-1185 .ISSN:1936-2625/IJCEP0013372